CLINICAL TRIAL: NCT01140672
Title: A Double Blind, 3rd Party Open, Placebo Controlled, Dose Escalating, Parallel Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of PF-04634817 In Healthy Volunteers
Brief Title: A Multiple Dose Study To Determine Safety, Tolerability, and Pharmacokinetics Of PF-04634817 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1261003
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Healthy volunteers; pharmacokinetics; safety; tolerability; multiple dosing; Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — PF-04634817

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cohort 1 (N=10) (Experimental): Placebo-controlled, multiple doses of PF-04634817 at 3 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817
- Cohort 2 (N=10) (Experimental): Placebo-controlled, multiple doses of PF-04634817 at 3 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817
- Cohort 3 (N=10) (Experimental): Placebo-controlled, multiple doses of PF-04634817 at 30 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817
- Cohort 4 (N=10) (Experimental): Placebo-controlled, multiple doses of PF-04634817 at 100 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817
- Cohort 5 (N=10) (Experimental): Placebo-controlled, multiple doses of PF-04634817 at 300 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817
- Cohort 6 (N=10) Optional cohort (Experimental): Placebo-controlled, multiple doses of PF-04634817 up to 300 mg per day for 14 days. (2 placebo: 8 active)
  Interventions: Drug: PF-04634817

INTERVENTIONS:
Drug: PF-04634817 — Oral solution of PF-04634817 at 3 mg will be given once daily for 14 days.
  Arms: Cohort 1 (N=10)
Drug: PF-04634817 — Oral solution of PF-04634817 at 3 mg will be given once daily for 14 days.
  Arms: Cohort 2 (N=10)
Drug: PF-04634817 — Oral solution of PF-04634817 at 30 mg will be given once daily for 14 days.
  Arms: Cohort 3 (N=10)
Drug: PF-04634817 — Oral solution of PF-04634817 at 100 mg will be given once daily for 14 days.
  Arms: Cohort 4 (N=10)
Drug: PF-04634817 — Oral solution of PF-04634817 at 300 mg will be given once daily for 14 days.
  Arms: Cohort 5 (N=10)
Drug: PF-04634817 — Cohort will only be dosed if necessary. Dose selected for this cohort may be a repeat of a previous cohort or intermediate dose not to exceed 300 mg.
  Arms: Cohort 6 (N=10) Optional cohort

SUMMARY:
The goals of this study are to evaluate the safety and tolerability of multiple ascending doses of PF-04634817 administered orally to healthy adult subjects. In additional, the plasma and urinary pharmacokinetics of multiple ascending doses of PF-04634817 administered orally to healthy adult subjects will be evaluated. Finally, the effect of multiple doses of PF-04634817 on circulating monocytes will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication;
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day;
* Nursing females;
* Females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, supine and standing vital sign measurements, 12-lead ECGs, blood and urine safety tests. | 14 days
Plasma PK Day 1: Cmax, Tmax, AUClast, AUCtau at all dose levels. Plasma PK Day 14: Cmax, Tmax, AUClast, AUCtau, AUCinf, t½, CL/F and Vss/F at all dose levels. | 14 days
AUCtau (Day 14) vs. AUCtau (Day 1) - estimate of accumulation ratio; Cmax (Day 14) vs. Cmax (Day 1); Tmax (Day 14) vs. Tmax (Day 1). | 14 days
Urinary PK: Aet (amount excreted in urine); Aet% at all doses of PF-04634817 where t = 24 hours on Day 1 and 14; CLr at all doses on Day 14. | 14 days
Pharmacodynamic: MCP-1 change from baseline. | 14 days

SECONDARY OUTCOMES:
Pharmacodynamic: p-ERK Inhibition in human monocytes: percent inhibition of monocyte p-ERK activity relative to the pre-dose baseline value | 14 days
MIP-1β stimulated CCR5 receptor internalization: percent inhibition of internalization relative to the pre-dose baseline value | 14 days
Absolute and percent change in circulating monocytes; Absolute and percent change in CD14+CD16+ monocytes. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261003&StudyName=A%20Multiple%20Dose%20Study%20To%20Determine%20Safety%2C%20Tolerability%2C%20and%20Pharmacokinetics%20Of%20PF-04634817%20In%20Healthy%20Adult%20Subjects